CLINICAL TRIAL: NCT01927315
Title: Effects of Fenofibrate on Endothelial Progenitor Cell Levels in Diabetic Patients With Retinopathy. A Randomized Controlled Trial.
Brief Title: Effects of Fenofibrate on Endothelial Progenitor Cells in Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2871P
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: Stem cells; Regeneration; Angiogenesis; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate (Experimental): Fenofibrate 145 mg (Fulcrosupra) oral tablets daily for 12 weeks
  Interventions: Drug: Fenofibrate 145 mg
- Placebo (Placebo Comparator): Placebo oral tablets daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate 145 mg — Tablets of Fulcrosupra 145 mg to be taken at 8.00 am daily for 12 weeks.
  Other Names: Fulcrosupra 145 mg
  Arms: Fenofibrate
Drug: Placebo — Oral Placebo tablets once daily
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
Long-standing diabetes is often complicated by retinopathy. The mechanisms that induce the development of diabetic retinopathy are incompletely understood and include alterations in bone marrow derived vasculogenic cells called "endothelial progenitor cells".

Fenofibrate is a PPAR-alpha agonist used for the treatment of mixed dislipidemia and hypertriglyceridemia. In a trial conducted in type 2 diabetic patients, the drug fenofibrate has reduced retinopathy-related endpoints suggesting a direct effect of the drug on the mechanisms that drive the development of this complication.

Herein, the investigators hypothesize that fenofibrate treatment can increase circulating EPC levels in diabetic patients with retinopathy, compared to placebo.

DETAILED DESCRIPTION:
Long-standing diabetes is often complicated by retinopathy. The mechanisms that induce the development of diabetic retinopathy are incompletely understood and include alterations in bone marrow derived vasculogenic cells called "endothelial progenitor cells".

Fenofibrate is a PPAR-alpha agonist used for the treatment of mixed dislipidemia and hypertriglyceridemia. In addition to lowering triglyceride-rich lipoproteins, PPAR-alpha agonism with fenofibrate has several additional molecular benefit on the vessel wall, such as reduction of inflammation. In a trial conducted in type 2 diabetic patients, the drug fenofibrate has reduced retinopathy-related endpoints suggesting a direct effect of the drug on the mechanisms that drive the development of this complication.

Preliminary data of ours on the effects of fenofibrate on cultured EPC show that this drug has the potential to improve EPC and, consequently, may benefit patients with retinopathy.

Herein, the investigators hypothesize that fenofibrate treatment can increase circulating EPC levels in diabetic patients with retinopathy, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* Diabetic retinopathy
* Age 18-70
* Both sexes

Exclusion Criteria:

* Age <18 or >70 at enrollment
* Hereditary muscle disorders
* Uncontrolled hypothyroidism
* Elevated alcohol consumption
* Renal failure
* Hepatic failure
* Allergy to fenofibrate or excipients
* Acute / chronic pancreatitis
* Pregnancy and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Endothelial progenitor cells | 12 weeks
  Change in endothelial progenitor cell (EPC) levels in fenofibrate-treated vs placebo-treated patients over 12 weeks.
Circulating progenitor cells | 12 weeks
  Change in circulating progenitor cell (CPC) levels in fenofibrate-treated vs placebo-treated patients over 12 weeks.

SECONDARY OUTCOMES:
Triglycerides | 12 weeks
  Change in Triglycerideslevels in fenofibrate-treated vs placebo-treated patients over 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Fadini, MD PhD, Principal Investigator — University of Padova
Locations (1):
- University Hospital of Padova, Diabetes Outpatient Clinic, Padua, Italy

REFERENCES:
- [Derived] Bonora BM, Albiero M, Morieri ML, Cappellari R, Amendolagine FI, Mazzucato M, Zambon A, Iori E, Avogaro A, Fadini GP. Fenofibrate increases circulating haematopoietic stem cells in people with diabetic retinopathy: a randomised, placebo-controlled trial. Diabetologia. 2021 Oct;64(10):2334-2344. doi: 10.1007/s00125-021-05532-1. Epub 2021 Aug 9. PMID 34368894